CLINICAL TRIAL: NCT00606892
Title: Varenicline Attenuates Some of the Subjective and Physiological Effects of Intravenous Nicotine in Humans.
Brief Title: Varenicline and Nicotine Interactions in Humans (VA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HIC # 0702002338; MIRECC 000000000 (Registry Identifier: Department of Veteran's Affairs); DPMC (Other: NIDA); R01DA014537 (NIH)
Record Dates: First submitted 2008-01-23; First posted 2008-02-05 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Smoking Cessation
Keywords: therapeutic effects
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Sugars; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo First, varenicline, + IV Nic (Experimental): Subjects received a Placebo tablet once per day for 4 days and then received a laboratory session where they were given ascending doses of Nicotine (0.1, 0.4, and 0.7 mg per 70 kg).After a minimum of a 5 day washout subjects then received varenicline tablet (1mg). once per day for 4 days and then received a laboratory session where they were given ascending doses of Nicotine (0.1,0.4,0.7 mg per 70kg).
  Interventions: Drug: Varenicline; Drug: Placebo; Drug: IV Nic
- Varenicline first, placebo, + IV Nic (Experimental): Subjects received Varenicline tablet (1 mg) per day for 4 days and then received a laboratory session where they were given ascending doses of Nicotine (0.1, 0.4, and 0.7 mg per 70 kg). After a washout of a minimum of 5 days subjects then received placebo tablet for per day for 4 days and then received a laboratory session where they were given ascending doses of Nicotine (0.1,0.4,, and 0.7mg per 70 kg).
  Interventions: Drug: Varenicline; Drug: Placebo; Drug: IV Nic

INTERVENTIONS:
Drug: Varenicline — Varenicline (1 mg per day) given for 4 days prior to laboratory session
  Other Names: Chantix
Drug: Placebo — Sugar Pill
  Other Names: Sugar Pill
Drug: IV Nic — IV Nicotine given during the laboratory session following 4 days of exposure to the study medication (varenicline or placebo). This nicotine was given during each laboratory session which followed the 4 days of exposure to either placebo then varenicline or varenicline then placebo.
  Other Names: IV Nicotine

SUMMARY:
To examine the effects of varenicline on the subjective, physiological and cognitive responses to intravenous nicotine. Varenicline is a partial nicotine agonist and it is approved as a treatment for smoking cessation. We predict that varenicline treatment will modify subjective, physiological and cognitive responses to IV nicotine.

DETAILED DESCRIPTION:
This will be a 2-4 week double-blind, placebo-controlled study. Twenty four male and female smokers will have two 4-day treatment periods, in which they will be randomized to varenicline (1 mg/day) or placebo. During the first 3 days of each treatment period, smokers will have daily clinic visits and receive their study medication. On Day 4, subjects will come to the laboratory, where they will receive ascending doses of intravenous (IV) nicotine (0.1, 0.4, and 0.7 mg per 70kg). This procedure will allow accurate assessment of varenicline effects on the subjective, physiological and cognitive responses to nicotine. Following a washout period, subjects will be crossed over to the alternative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 55 years
* History of smoking daily for the past 12 months, at least 15 cigarettes daily
* Carbon Monoxide (Alveolar) level > 10ppm
* For women: not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods

Exclusion Criteria:

* History of heart disease, renal or hepatic diseases
* other medical conditions that the physician investigator deems as contraindicated for the subject to be in the study
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* recent psychiatric diagnosis and treatment for Axis I disorders including
* major depression, bipolar affective disorder,
* schizophrenia and panic disorder within the past year
* Current dependence on alcohol
* drugs or treatments for drug
* alcohol addiction within the past 5 years
* Allergy to varenicline

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University Associate Professor
Locations (1):
- Veterans Affairs Hospital, West Haven, Connecticut, United States

REFERENCES:
- [Result] Sofuoglu M, Herman AI, Mooney M, Waters AJ. Varenicline attenuates some of the subjective and physiological effects of intravenous nicotine in humans. Psychopharmacology (Berl). 2009 Nov;207(1):153-62. doi: 10.1007/s00213-009-1643-z. Epub 2009 Aug 20. PMID 19693492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the New Haven Connecticut area through newspaper advertisements and fliers from the summer of 2007 thru the winter of 2008.
Pre-assignment Details: There was no special pre-assignment procedures for this study. Thirty seven smokers signed a consent form with only 17 randomized. 13 smokers never return to clinic after signing a consent form. 2 smokers were excluded secondary to poor IV access. 5 smokers had dropped out due to a scheduling conflict.
Groups:
- Placebo First, Then Varenicline: Subject received a placebo tablet once per day for 4 days and then received a laboratory session where they were given ascending dose of Nicotine (0.1,0.4, and 0.7mg per70kg). After a minimum washout period of 5 days,then subjects received Varenicline (1mg) per day for 4 days and then received a laboratory session where they were given ascending doses of Nicotine (0.1, 0.4, and 0.7mg per 70kg).
- Varenicline First, Then Placebo: Subjects received Varenicline (1mg) per day for 4 days and then received a laboratory session where they were given ascending doses of Nicotine (0.1, 0.4, and 0.7mg per 70kg).After a minimum of washout period of 5 days, then subjects received a placebo tablet once per day for 4 days and then received a laboratory session where they were given ascending dose of Nicotine (0.1,0.4, and 0.7mg per70kg).
Period: Adaptation
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: First Intervention
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 9 | 8
Completed | 8 | 4
Not Completed | 1 | 4
Not completed — Protocol Violation | 1 | 4
Period: Washout Period
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Varenicline | Varenicline First, Then Placebo
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 37 subjects signed consent. 17 subjects received the first treatment. Five subjects dropped out due to non-compliance with study procedures prior to study completion, and therefore were not included in the analysis. The 12 subjects who completed both interventions were included in the analysis.
Groups:
- Entire Study Population: Includes all subjects who completed the study. (The total number of subjects who were enrolled in both arms of the study.)
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Secondary Outcome: Mean Reaction Time (RT) on Modified Stroop Task.
Description: A Modified stroop task was used to assess attentional responses to smoking and negative affect cues. Cues were presented as blue, red or green text. Subjects completed 2 counterbalanced blocks (60 trials per block). One block contained smoking cues and neutral cues. The other block contained negative affect cues and a different set of matched neutral cues. The 2 blocks were administered twice during each experimental session - prior to nicotine infusion, and 30 mins after the last nicotine infusion (2 hrs and 45 mins after medication dosing). The Stroop effect is a differential RT when identifying the colors of words presented as neutral cues vs. emotional cues (i.e. smoking or negative affect cues).
Time Frame: pre-nicotine, and 30 min after last nicotine infusion (Post-Nicotine)
Population: Data from all subjects who completed both experimental sessions (nicotine infusion after 4 days of placebo and also 4 days of varneicline, n=12) are presented. RT's < 100 ms, or > 1501 ms were excluded from the analysis (>3 SD's of the mean). The data presented are the mean RT's to identifying word colors under each treatment condition.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Placebo, Pre-Nicotine: Mean reaction time during modified Stroop task under the placebo condition and prior to the nicotine infusions.
- Placebo, Post-Nicotine: Mean reaction time during modified Stroop task under the placebo condition and 30 minutes after the nicotine infusions.
- Varenicline, Pre-Nicotine: Mean reaction time during modified Stroop task under the varenicline condition prior to the nicotine infusions.
- Varenicline, Post-Nicotine: Mean reaction time during modified Stroop task under the varenicline condition and 30 minutes after the nicotine infusions.
Arm/Group | Placebo, Pre-Nicotine | Placebo, Post-Nicotine | Varenicline, Pre-Nicotine | Varenicline, Post-Nicotine
Number analyzed (Participants) | 12 | 12 | 12 | 12
milliseconds
  Smoking Block | 722.3 (131.3) | 693.1 (129.4) | 660.1 (137.8) | 624.2 (100.1)
  Neutral Block- Smoking Cue | 702.3 (148.6) | 686.7 (134.1) | 652.1 (115.5) | 618.6 (104.7)
  Negative Affect block | 679.0 (104.1) | 641.3 (114.9) | 665.8 (177.1) | 631.7 (128.6)
  Neutral Block- Negative Affect Cue | 692.5 (117.5) | 661.5 (111.1) | 644.8 (122.8) | 618.6 (108.5)
Statistical Analysis 1: Comparison: Placebo, Pre-Nicotine vs Placebo, Post-Nicotine vs Varenicline, Pre-Nicotine vs Varenicline, Post-Nicotine; A mixed-effect repeated-measures crossover model with fixed main effect terms of treatment (placebo or varenicline) and time of measurement (Pre-Nicotine or Post-Nicotine) was utilized. Interactions between main effect terms were also analyzed; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — Significant treatment or treatment-by-time interactions were followed up by post hoc comparisons of placebo vs. varenicline for time (Pre- vs. Post-Nicotine infusion) and testing block (Smoking Block vs. Negative Affect Block)

2. Secondary Outcome: Cotinine Levels
Description: Subject Cotinine Levels before each laboratory session.
Time Frame: Before each laboratory session on day 5
Population: Subjects finishing the complete study. (n=12)
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo: The mean cotinine levels for subjects under the placebo condition.
- Varenicline (1 mg): The mean cotinine levels for subjects under the varenicline condition.
Arm/Group | Placebo | Varenicline (1 mg)
Number analyzed (Participants) | 12 | 12
ng/mL | 202 (41) | 185 (38)
Statistical Analysis 1: Comparison: Placebo vs Varenicline (1 mg); Test type: Superiority or Other; p < 0.3, ANOVA; F(1,10)=1.1; Mean Difference (Final Values) = 17, Standard Deviation 40

3. Primary Outcome: Subjective Responses to Intravenous Nicotine
Description: The Drug Effects Questionaire( DEQ) is a 7-item psychometric that measures the following subjective categories: 'drug strength',' high', 'feels stimulated', 'good effects', 'bad effects', 'head rush', and 'like the drug'. Smokers rated each item on a 100 millimeter scale from "not at all" (a score of 0) to "extremely" with a maximum score of 100.
Time Frame: 30 minutes after each nicotine infusion
Population: All participants who complete all interventions.
Measure: Mean (Standard Error); unit: millimeters
Groups:
- Placebo/ Low Dose Nictoine: The average peak change (change score) in the subjective responses to the 7-items of the DEQ to the low dose (0.1) of IV nicotine under the placebo condition.
- Placebo/ Medium Dose Nicotine: The average peak change (change score) in the subjective responses to the 7-items of the DEQ to the medium dose (0.4) of IV nicotine under the placebo condition.
- Placebo/High Dose Nicotine: The average peak change (change score) in the subjective responses to the 7-items of the DEQ to the high dose (0.7) of IV nicotine under the placebo condition.
- Varenicline/ Low Dose Nicotine: The average peak change (change score) in the subjective responses to the 7-items of the DEQ to the low dose (0.1) of IV nicotine under the varenicline condition.
- Varenicline/ Medium Dose Nicotine: The average peak change (change score) in the subjective responses to the 7-items of the DEQ to the medium dose (0.4) of IV nicotine under the varenicline condition.
- Varenicline/ High Dose Nicotine: The average peak change (change score) in the subjective responses to the 7-items of the DEQ to the high dose (0.7) of IV nicotine under the varenicline condition.
Arm/Group | Placebo/ Low Dose Nictoine | Placebo/ Medium Dose Nicotine | Placebo/High Dose Nicotine | Varenicline/ Low Dose Nicotine | Varenicline/ Medium Dose Nicotine | Varenicline/ High Dose Nicotine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
millimeters
  High | 23 (8) | 38 (10) | 51 (10) | 14 (4) | 27 (7) | 37 (8)
  Head Rush | 24 (8) | 40 (9) | 51 (9) | 11 (4) | 28 (7) | 37 (8)
  Feels Stimulated | 25 (8) | 34 (10) | 38 (10) | 11 (4) | 24 (8) | 35 (9)
  Drug Strength | 24 (8) | 41 (9) | 58 (09) | 16 (4) | 32 (7) | 40 (8)
  Bad Effects | 7 (3) | 15 (7) | 23 (8) | 8 (3) | 8 (3) | 20 (8)
  Good Effects | 19 (8) | 30 (8) | 45 (10) | 22 (8) | 25 (8) | 34 (9)
  Like the Drug | 18 (8) | 27 (9) | 35 (10) | 14 (4) | 25 (8) | 35 (9)
Statistical Analysis 1: Comparison: Placebo/ Low Dose Nictoine vs Placebo/ Medium Dose Nicotine vs Placebo/High Dose Nicotine vs Varenicline/ Low Dose Nicotine vs Varenicline/ Medium Dose Nicotine vs Varenicline/ High Dose Nicotine; A mixed-effect repeated-measures crossover model including fixed main effects for treatment condition (placebo or varenicline), time of measurement and interactions between treatment and time, was utilized. Because multiple measurements were collected before and after each nicotine dose, a change score (maximum post dose score - pre dose baseline) was used in the analysis; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — Values of p<0.05 were considered statistically significant, based on 2-tailed tests. Significant treatment, or treatment-by-time interactions were followed by post hoc comparisons. To account for multiple testing, significance was set at p<0.016; Mean Difference (Final Values) = 0

4. Secondary Outcome: Heart Rate
Description: The average peak change (change score = maximum post dose score minus predose baseline) in heart rate was calculated.
Time Frame: 30 minutes after each nicotine infusion
Population: Changes in heart rate, systolic and diastolic blood pressure during the experimental sessions were analyzed on all subjects who completed both experimental sessions (n=12).
Measure: Mean (Standard Error); unit: beats per minute
Groups:
- Placebo / Low Dose Nicotine: The average peak change (change score) in heart rate after nicotine (0.1mg per70kg) infusion under the placebo condition.
- Placebo/ Medium Dose Nicotine: The average peak change (change score) in heart rate after nicotine (0.4mg per 70kg) infusion under the placebo condition.
- Placebo/High Dose Nicotine: The average peak change (change score) in heart rate after nicotine (0.7mg per 70kg) infusion under the placebo condition.
- Varenicline/ Low Dose Nicotine: The average peak change (change score) in heart rate after nicotine (0.1mg per 70kg) infusion under the varenicline condition.
- Varenicline/ Medium Dose Nicotine: The average peak change (change score) in heart rate after nicotine (0.4mg per 70kg) infusion under the varenicline condition.
- Varenicline / High Dose Nicotine: The average peak change (change score) in heart rate after nicotine (0.7mg per 70kg) infusion under the varenicline condition.
Arm/Group | Placebo / Low Dose Nicotine | Placebo/ Medium Dose Nicotine | Placebo/High Dose Nicotine | Varenicline/ Low Dose Nicotine | Varenicline/ Medium Dose Nicotine | Varenicline / High Dose Nicotine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
beats per minute | 7 (1) | 13 (2) | 16 (2) | 2 (2) | 5 (1) | 5 (2)
Statistical Analysis 1: Comparison: Placebo / Low Dose Nicotine vs Placebo/ Medium Dose Nicotine vs Placebo/High Dose Nicotine vs Varenicline/ Low Dose Nicotine vs Varenicline/ Medium Dose Nicotine vs Varenicline / High Dose Nicotine; A mixed-effect, repeated-measures, crossover model was used with fixed main effects for treatment (placebo or varenicline), and time after treatment. Interactions between main effects were also analyzed; Test type: Superiority or Other; p < 0.05, ANOVA — Post hoc comparisons of effects of varenicline versus placebo for different nicotine doses were performed and significance was adjusted for multiple testing using a p value of P<0.016; Two-tailed tests were applied for main effects with P<0.05

5. Secondary Outcome: Changes in Systolic and Diastolic Blood Pressure
Description: The average peak change (change score = maximum post dose score minus predose baseline) in systolic and diastolic blood pressure after nicotine infusion.
Time Frame: 30 minutes after each nicotine infusion
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Placebo / Low Dose Nicotine: The average peak change (change score) in systolic and diastolic blood pressure after nicotine (0.1mg per 70kg) infusion under the placebo condition.
- Placebo/ Medium Dose Nicotine: The average peak change (change score) in systolic and diastolic blood pressure after nicotine (0.4mg per 70kg) infusion under the placebo condition.
- Placebo/High Dose Nicotine: The average peak change (change score) in systolic and diastolic blood pressure after nicotine (0.7mg per 70kg) infusion under the placebo condition.
- Varenicline/ Low Dose Nicotine: The average peak change (change score) in systolic and diastolic blood pressure after nicotine (0.1mg per 70kg) infusion under the varenicline condition.
- Varenicline/ Medium Dose Nicotine: The average peak change (change score) in systolic and diastolic blood pressure after nicotine (0.4mg per 70kg) infusion under the varenicline condition.
- Varenicline / High Dose Nicotine: The average peak change (change score) in systolic and diastolic blood pressure after nicotine (0.7mg per 70kg) infusion under the varenicline condition.
Arm/Group | Placebo / Low Dose Nicotine | Placebo/ Medium Dose Nicotine | Placebo/High Dose Nicotine | Varenicline/ Low Dose Nicotine | Varenicline/ Medium Dose Nicotine | Varenicline / High Dose Nicotine
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
mm Hg
  Systolic Blood Pressure | 12 (4) | 16 (2) | 8 (3) | 7 (2) | 13 (3) | 16 (3)
  Diastolic Blood Pressure | 7 (2) | 6 (2) | 5 (1) | 5 (2) | 6 (2) | 7 (2)

ADVERSE EVENTS:
Groups:
- Placebo First, Then Varenicline, First Intervention: Subjects received a placebo tablet once per day for 4 days prior to the first laboratory session (first intervention) where they were given ascending doses of Nicotine (0.1, 0.7mg per 70kg).
- Varenicline First, Then Placebo, First Intervention: Subjects received varenicline once per day for 4 days prior to the first laboratory session (first intervention) where they were given ascending doses of Nicotine (0.1, 0.7mg per 70kg).
- Adaptation - Placebo First, Then Varenicline: Subjects randomized to the 'Placebo first' condition participated in a laboratory session where they were given ascending doses of Nicotine (0.1, 0.4, 0.7mg per 70 kg) to assess tolerability prior to the study medication intervention.
- Adaptation - Varenicline First, Then Placebo: Subjects randomized to the 'Varenicline first' condition first received a laboratory session where they were given ascending doses of Nicotine (0.1, 0.4, 0.7mg per 70 kg) to assess tolerability before receiving the study medication.
- Placebo First, Then Varenicline, Second Intervention: Subjects crossed-over from the first intervention and received varenicline once per day for 4 days prior to the second laboratory session (second intervention) where they were given ascending doses of Nicotine (0.1, 0.7mg per 70kg).
- Varenicline First, Then Placebo, Second Intervention: Subjects crossed-over from the first intervention (varenicline) and received placebo once per day for 4 days prior to the second laboratory session (second intervention) where they were given ascending doses of Nicotine (0.1, 0.7mg per 70kg).
Arm/Group | Placebo First, Then Varenicline, First Intervention | Varenicline First, Then Placebo, First Intervention | Adaptation - Placebo First, Then Varenicline | Adaptation - Varenicline First, Then Placebo | Placebo First, Then Varenicline, Second Intervention | Varenicline First, Then Placebo, Second Intervention
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/8 | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No